CLINICAL TRIAL: NCT04730856
Title: Standard vs High Prophylactic Doses or Anticoagulation in Patients With High Risk of Thrombosis Admitted With COVID-19 Pneumonia (PROTHROMCOVID)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTHROMCOVID
Record Dates: First submitted 2021-01-14; First posted 2021-01-29 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Thrombosis
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tinzaparin 4500 UI/day (Active Comparator): Procedure: Tinzaparin 4500 UI/day SC until hospital discharge.
  Interventions: Drug: Tinzaparin
- Tinzaparin 100 UI/Kg/day (Active Comparator): Procedure: Tinzaparin 100 UI/Kg/day SC until hospital discharge.
  Interventions: Drug: Tinzaparin
- Tinzaparin 175 UI/Kg/day (Active Comparator): Procedure: Tinzaparin 175 UI/Kg/day SC until hospital discharge.
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — day subcutaneously • Follow-up phase 1 (Day 15 to day 30): The information is obtained at discharge and on day +14, + 28 on 30 days. The latter information is obtained from patients, from medical records or by telephone contact at the patient's home.
  • Follow-up phase 2 (At 3 months: Information is obtained from patients, medical records, or by telephone contact at the patient's home.

SUMMARY:
The main objective is to evaluate the efficacy and safety of three doses of tinzaparin (prophylactic, intermediate and therapeutic) in hospitalized patients with COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to hospital with COVID-19, PCR and/or Antigens Test + SARS-CoV-2 infection or (presence of infiltrate compatible with Chest X-ray or TC)
2. Patients with, at least, one of the following evolution disease risk criteria:

   * Sat 02<94%
   * Need for oxygen therapy or pAO2/FiO2<300mmHg or estimated PaO2/FiO2 based on SpO2/FiO2<300 mmHg.
   * DD>1000µg/L
   * PCR >150mg/L
   * IL6 >40pg/ml
3. Age > 18 years
4. Weight 50-100 Kg
5. After receiving oral and written information about the study, patient must give Informed Consent duly signed and dated before performing any activity related to the study.

Exclusion Criteria:

1. Patients who need mechanical ventilation (invasive or non-invasive), high flow nasal cannula or admission to ICU at the moment of randomization.
2. Current diagnosis of acute bronchial asthma attack.
3. History or clinical suspicion of pulmonary fibrosis.
4. Current diagnosis or suspicion of pulmonary thromboembolism or deep vein thrombosis.
5. Patients who need anticoagulant treatment due to previous venous or arterial thrombotic disease, or due to atrial fibrillation.
6. Patients with pneumonectomy or lobectomy.
7. Renal failure with Glomerular filtration <30 ml/min/1.73m2
8. Patients with contraindication for anticoagulant treatment.
9. Congenital bleeding disorders.
10. Hypersensitivity to tinzaparin or UFH or some of its excipients.
11. History of heparin-induced thrombocytopenia.
12. Active bleeding or situation that predispose to bleeding.
13. Moderate or severe anaemia (Hb<10 g/dl)
14. Low platelet count < 80000/µl
15. Patients with life expectancy less than 3 months due to primary disease evaluated by the physician.
16. Patients currently intubated or intubated between the screening and the randomization.
17. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Combined variable that includes outcomes 2, 3 and 4 detailed below | 30 days
  Combined variable that includes outcomes 2, 3 and 4 detailed below (reduction of suspicion of systemic thrombotic symptomatic events and/or need for mechanical ventilation and/or death at day 30 after randomization).
Reduction of suspicion of systemic thrombotic symptomatic events | 30 days
  Reduction of symptomatic thrombotic events: rate of venous thromboembolism confirmed by objective test.
Use of Mechanical ventilation invasive or non invasive including high flow nasal cannula oxigen | 30 days
  Mechanical ventilation (invasive or non-invasive) free survival.
Overall survival at 30 days. | 30 days
  Overall survival at 30 days: number of deaths.

SECONDARY OUTCOMES:
Number of bleedings and adverse reactions | 90 days
  Safety of the different strategies of prophylaxis and anticoagulation: number of bleedings and adverse reactions in each group:
  Evaluation of the following variables:
  Incidence of major bleeding, defined as meeting any of these criteria:
  a) fatal bleeding or bleeding that occurs in a critical area or organ (for example, intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome), b ) causes a drop in hemoglobin level of 20 g/L or more, or c) requires the transfusion of 2 or more units of whole blood or packed red blood cells.
  Incidence of clinically relevant non-major bleeding: manifest, spontaneous or post-traumatic bleeding, which does not meet the criteria for major bleeding but which in the judgment of the investigator is relevant.
  Incidence of clinically relevant bleeding: all major and non-major hemorrhages clinically relevant.
  Incidence of adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Muñoz Rivas, Study Chair — Hospital Universitario Infanta Leonor
Locations (18):
- Spain (18):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario del Vinalopó, Alicante
  - Hospital Clínic Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - Hospital de Emergencias Enfermera Isabel Zendal, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro, Vigo

REFERENCES:
- [Background] Lew TW, Kwek TK, Tai D, Earnest A, Loo S, Singh K, Kwan KM, Chan Y, Yim CF, Bek SL, Kor AC, Yap WS, Chelliah YR, Lai YC, Goh SK. Acute respiratory distress syndrome in critically ill patients with severe acute respiratory syndrome. JAMA. 2003 Jul 16;290(3):374-80. doi: 10.1001/jama.290.3.374. PMID 12865379
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Derived] Munoz-Rivas N, Aibar J, Gabara-Xanco C, Trueba-Vicente A, Urbelz-Perez A, Gomez-Del Olmo V, Demelo-Rodriguez P, Rivera-Gallego A, Bosch-Nicolau P, Perez-Pinar M, Rios-Prego M, Madridano-Cobo O, Ramos-Alonso L, Alonso-Carrillo J, Francisco-Albelsa I, Marti-Saez E, Maestre-Peiro A, Mendez-Bailon M, Hernandez-Rivas JA, Torres-Macho J; PROTHROMCOVID Trial Investigators. Efficacy and Safety of Tinzaparin in Prophylactic, Intermediate and Therapeutic Doses in Non-Critically Ill Patients Hospitalized with COVID-19: The PROTHROMCOVID Randomized Controlled Trial. J Clin Med. 2022 Sep 24;11(19):5632. doi: 10.3390/jcm11195632. PMID 36233500